CLINICAL TRIAL: NCT02828644
Title: An Exploratory Study to Assess the Sustained Effects of Digital Therapy in Pediatric Subjects 8 to 12 Years Old With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Software Treatment for Actively Reducing Severity of ADHD - Follow Up
Acronym: STARS-ADHD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Akili-001R-FollowUp
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVO Multitasking (Active Comparator): EVO Multitasking is a digital intervention that requires subjects to navigate a character through a game-like space, while collecting objects, in a fixed period of time. The intervention was administered to the subjects during the parent study (Akili-001R)
  Interventions: Device: EVO
- EVO Words (Active Comparator): EVO Words is a digital intervention that requires subjects to spell as many words as possible, by connecting letters in a game-like grid, in a fixed period of time. The intervention was administered to the subjects during the parent study (Akili-001R)
  Interventions: Device: EVO

INTERVENTIONS:
Device: EVO — videogame-like digital therapy

SUMMARY:
This is an exploratory study to assess potential maintenance of clinical benefit (cognition and symptoms) following 4 weeks of at-home digital therapy in ADHD children.

DETAILED DESCRIPTION:
The study will be a blinded (investigators and outcome assessors), randomized (from parent study Akili-001R), parallel group, follow-up study of the sustained effects of 4-weeks of treatment with either AKL-T01 (EVO Multi) game-based digital therapy or AKL-T09 (EVO Words) game-based digital therapy.

The trial will consist of 4 visits: Screening (to be conducted at the same time as the end-of-study visit for the parent study Akili-001R), FU-Day 28 visit (conducted in clinic), and FU-Day 56 and FU-Day 84 visits (conducted remotely via electronically captured parent reported outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Completed Akili Study Akili-001R including all clinical assessments at DAY28 per the study protocol
* Ability to comply with all the testing and requirements per this protocol

Exclusion Criteria:

* Participant is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation or self-injurious behavior as measured by C-SSRS at screening
* Participant has demonstrated clinically significant deterioration in functioning as assessed by PI and other study staff that would contraindicate continued participation in the follow-up study

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kollins, PhD, Principal Investigator — Duke Clinical Research Institution
Locations (14):
- United States (14):
  - Melmed Center, Scottsdale, Arizona
  - Avida, Inc., Newport Beach, California
  - University of California Davis MIND Institute, Sacramento, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Meridien Research, Bradenton, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - South Shore Psychiatric Services, Marshfield, Massachusetts
  - Midwest Research Group, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - Duke Child and Family Study Center, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - The Neuropsychiatric Clinic at Carolina Partners, Raleigh, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- AKL-T01 (EVO Multi): AKL-T01, or EVO Multi, is a digital intervention that requires subjects to navigate a character through a game-like space, while collecting objects, in a fixed period of time. The intervention was administered to the subjects during the parent study (Akili-001R, NCT02674633)
- AKL-T09 (EVO Words): AKL-T09, or EVO Words, is a digital intervention that requires subjects to spell as many words as possible, by connecting letters in a game-like grid, in a fixed period of time. The intervention was administered to the subjects during the parent study (Akili-001R, NCT02674633)
Period: Overall Study
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Started | 88 | 87
Completed | 65 | 65
Not Completed | 23 | 22
Not completed — Lost to Follow-up | 23 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words) | Total
Number analyzed (Participants) | 88 | 87 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 88 | 87 | 175
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 21 | 51
  Male | 58 | 66 | 124
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88 | 87 | 175

OUTCOME MEASURES:

1. Primary Outcome: Sustained Effects in Attention From End-of-treatment (Follow-Up Day 0) to Follow-Up Day 28 Within Groups That Were Previously Randomized to Receive 4 Weeks of Digital Therapy
Description: TOVA API is a comparison of the subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated. The API is calculated from variability, response time, and d' (D Prime) using the following formula:
  API = Response Time Z score (Half 1) + d' Z score (Half 2) + Variability Z score (Total) + 1.80
  where Response Time is the average time it takes to respond correctly to a target, d' score is a response discriminability score reflecting the ratio of hits to "false alarms", and Variability is a measure of consistency of speed of responding based on the standard deviation of the mean correct response times. API tells how similar the score is to the ADHD profile. A score of less than 0 indicates that the subject had similar performance to a normative ADHD population. A lower score indicates a more severe ADHD profile.
  The calculation for difference in TOVA API was API at Day 28 minus API at Day 0 of this study.
Time Frame: Day 0 to Day 28
Population: All subjects who were randomized to the AKL-T01 arm in 001R/NCT02674633, completed 4 weeks of at-home play, and completed the Day 0 and Day 28 visits of this study.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | AKL-T01 (EVO Multi)
Number analyzed (Participants) | 65
z-score | -0.407 (2.823)

2. Secondary Outcome: Sustained Effects in Attention From End-of-treatment (Follow-Up Day 0) to Follow-Up Day 28 Across Groups That Were Previously Randomized to Receive 4 Weeks of Digital Therapy
Description: as for outcome 1
Time Frame: Day 0 to Day 28
Population: All subjects who were enrolled in 001R/NCT02674633, completed 4 weeks of at-home play, and completed the Day 0 and Day 28 visits of this study.
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- AKL-T01 (EVO Multi): EVO Multitasking is a digital intervention that requires subjects to navigate a character through a game-like space, while collecting objects, in a fixed period of time. The intervention was administered to the subjects during the parent study (Akili-001R, NCT02674633)
- AKL-T09 (EVO Words): EVO Words is a digital intervention that requires subjects to spell as many words as possible, by connecting letters in a game-like grid, in a fixed period of time. The intervention was administered to the subjects during the parent study (Akili-001R, NCT02674633)
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
Number analyzed (Participants) | 65 | 65
z-score | -0.407 (2.823) | -0.615 (3.338)

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | AKL-T01 (EVO Multi) | AKL-T09 (EVO Words)
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/87
Other Adverse Events (participants affected / at risk) | 0/88 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT02828644/Prot_SAP_000.pdf